CLINICAL TRIAL: NCT01163786
Title: A Phase 2 Proposal to Test the Efficacy and Tolerability of Bortezomib in Pulmonary Chronic GVHD
Brief Title: A Proposal to Test the Efficacy and Tolerability of Bortezomib in Pulmonary Chronic GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed due to low accrual before the accrual goal was reached
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 09H7; NU 09H7 (Other: Northwestern University Cancer Center); STU00022160 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-07-07; First posted 2010-07-16 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Bronchiolitis Obliterans
Keywords: Bortezomib GVHD Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): Patients will Receive 2 4week cycles of Bortezomib. Each cycle will consist of weekly bortezomib with a 2 week interval between cycles.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Each patient will receive 2 cycles of Bortezomib. For each cycle Bortezomib wil be given once a week, 1.3mg/m2 for 4 weeks with 2 weeks between each cycle.
  Other Names: Velcade

SUMMARY:
Approximately 10,000 allogeneic hematopoietic stem cell transplants (HSCT) are performed annually in the US for various indications. Bronchiolitis obliterans (BO) is the most common late noninfectious complication following allogeneic hematopoietic stem cell transplant. Prognosis of BO in the allogeneic HSCT setting is dismal and there are no therapies proven to be consistently effective. The exact incidence is not clear but may be as high as 30%2 . Risk factors include new or ongoing chronic graft versus host disease (cGVHD), age, antecedent obstructive airways disease and viral infections1. BO is characterized physiologically by progressive irreversible airflow obstruction and pathologically by luminal occlusion of the distal airways due to progressive scarring3. The pathogenesis is not completely understood but the cytokine transforming growth factor-beta 1 (TGF-b1), important for both tissue repair and fibrosis, is thought to play a pivotal role. Bortezomib, an FDA approved proteasomal inhibitor inhibits TGF-b1 signaling in vitro and protects against lung injury/fibrosis in bleomycin mouse model as well as in a mouse model for skin fibrosis. This is consistent with other data in the literature that proteasomal inhibition can prevent the development of fibrosis. Thus the investigators propose to test the safety, tolerability and efficacy of bortezomib in chronic pulmonary GVHD (BO).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Day >100 after allogeneic hematopoietic stem cell transplantation
* Underlying cancer in remission
* Decrease in FEV1 of ≥12% from the pre-transplant baseline (FEV1/FVC ratio <0.8)
* No evidence of acute infection
* ANC >1000
* Platelets >50,000
* Age 18-70
* ECOG performance Status 0-2.

Exclusion Criteria:

* Patient has a platelet count of less than 50,000 within 14 days before enrollment.
* Patient has an absolute neutrophil count of less 1000 within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of < 20 ml/minute within 14 days before enrollment.
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum b-human chorionic gonadotropin (b-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Inability of give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manu Jain, MD, MS, Principal Investigator — Northwestern University; Jayesh Mehta, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on July 20, 2010 with an accrual goal of up to 20 evaluable patients. The first patient being enrolled on the study on October 7th 2010. The study was closed permanently on August 31 2015 before the accrual goal was met with 17 patients being treated on study.
Pre-assignment Details: Patients were diagnosed with pulmonary Chronic Graft Verses Host Disease (p-CGVHD) after having undergone allogeneic hematopoietic stem cell transplant (HSCT). Patients were required to be less than 100 days post HSCT, with an absolute decrease of 12% or more in forced expiratory volume in 1 second (FEV1) from pre-transplant baseline.
Groups:
- Bortezomib: Patients will receive 2 cycles of Bortezomib (given weekly for 4 weeks) for a total of 8 doses of Bortezomib. Each cycle will consist of weekly bortezomib with a 2 week interval between cycles.
  Bortezomib: Each patient will receive 2 cycles of Bortezomib. For each cycle Bortezomib will be given once a week, 1.3mg/m2 for 4 weeks with 2 weeks between each cycle.
Period: Treatment With Bortezomib
Arm/Group | Bortezomib
Started | 17
Completed 1st Cycle | 17
Completed 2nd Cycle | 14 (One patient completed cycle 2 but missed one dose of Bortezomib.)
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Period: Completed Follow up (Visit 9 and 10)
Arm/Group | Bortezomib
Started | 14
Completed Week 12 Follow up (Visit 9) | 14
Completed Week 18 Follow up (Visit 10) | 13
Completed | 13
Not Completed | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Disease [Count of Participants; unit: Participants]
  Acute Leukemia | 6
  Chronic Myelogenous Leukemia | 3
  Lymophoma | 4
  Myeloma | 2
  Other | 2
Sex Matching of Transplantation [Count of Participants; unit: Participants]
  Female-female | 1
  Female-male | 3
  male-female | 5
  male-male | 8
Transplant Type [Count of Participants; unit: Participants]
  Matched Sibling | 12
  Matched unrelated | 4
  Mini matched unrelated | 1
Plumonary Function Testing (PFT) at time of transplant [Mean (Standard Deviation); unit: percentage]
  Forced Expiratory Volume in 1 Second (FEV1) | 90 (17)
  Forced Vital Capacity (FVC) | 89 (18)
  FEV/FVC | 81 (5)
lumonary Function Testing at time of pulmonary Chronic Graft-verses-host disease (pGVHD) Diagnosis [Mean (Standard Deviation); unit: percentage]
  Forced Expiratory Volume in 1 Second (FEV1) | 47 (16)
  Forced Vital Capacity (FVC) | 60 (15)
  FEV/FVC | 61 (14)
Time from transplant to pGVHD diagnosis [Mean (Standard Deviation); unit: years] | 3.36 (1.88)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Function as Measured by Forced Expiratory Volume in 1 Second (FEV1) Decline
Description: FEV1 will be measured by spirometry assessments at baseline (pre-transplant baseline - prior to pulmonary chronic graft-versus-host disease (p-CGVHD)) during treatment (10 weeks) and at follow up visit 9 (at 12 weeks) and at follow up visit 10 (at 18 weeks) with patients having spirometry tested up to 6 times from screening to the end of the study. FEV1 is reported as slopes computed by dividing difference in FEV1 by time in months.
Time Frame: Mean time to diagnosis (from transplant to p-CGVHD ) of 3.36 years (+/- 1.88 years) and up to 18 weeks after baseline
Measure: Median (Full Range); unit: percentage per month
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
percentage per month
  Prior to diagnosis of p-CGVHD | -1.06 [-5.36 to -0.33]
  During Treatment with Bortezomib | -0.25 [-9.42 to 3.52]

2. Secondary Outcome: Exercise Tolerance- 6 Minute Walk
Description: Patients will have an exercise tolerance assessment defined as a 6 minute walk completed at cycle 1 (week 1) and cycle 2 (week 5) of treatment and visit 9 (12 weeks) and visit 10 (18 weeks).
Time Frame: Up to 18 weeks from baseline
Population: Data was collected but not analyzed due to the study closing before accrual was met. Below is data on how many patients started 6 minute walk and how many patients stopped before reaching 6 minutes at each time point is shown below.
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 13
participants
  Cycle 1 (Visit 1): Started 6 Minute walk | 13
  Cycle 1 (Visit 1): Stopped before 6 minutes | 3
  Cycle 1(Visit 1):Declined walk | 0
  Cycle 2 (Visit 5) : Started 6 Minute walk: number analyzed (Participants) | 3
  Cycle 2 (Visit 5) : Started 6 Minute walk | 3
  Cycle 2 (Visit 5) : Stopped before 6 minutes | 0
  Cycle 2(Visit 5):Declined walk | 0
  Follow up/Visit 9: Started 6 Minute walk: number analyzed (Participants) | 7
  Follow up/Visit 9: Started 6 Minute walk | 6
  Follow up/Visit 9 : Stopped before 6 minutes | 1
  Follow up/Visit 9: Declined walk | 1
  Follow up/Visit 10 : Started 6 Minute walk: number analyzed (Participants) | 6
  Follow up/Visit 10 : Started 6 Minute walk | 5
  Follow up/Visit 10 : Stopped before 6 minutes | 1
  Follow up/Visit 10: Declined walk | 1

3. Secondary Outcome: Short Form (SF)-36 Health Survey
Description: This is a quality of life questionnaire which yields scores for 8 domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health). This questionnaire will be completed by patients on Visit 1 (week 1), Visit 5 (week 5), Visit 8 (week 8), Visit 9 (12 weeks), and Visit 10 (18 weeks).
  Questionnaires were scored per the scoring rules for the RAND 36-Item Health Survey (version 1.0) A high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Time Frame: up to 18 weeks
Population: Data was collected but not analyzed. Averages for each patient at each timepoint are shown below. N/a is shown for timepoints where data was not collected.
Measure: Number; unit: Average Score
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
Average Score
  Pt #01 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #01 Physical Functioning : Visit 1 | 30
  Pt #01 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #01 Physical Functioning : Visit 5 | 55
  Pt #01 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #01 Physical Functioning : Visit 8 | NA — Data not collected
  Pt #01 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #01 Physical Functioning : Visit 9 | NA — Data not collected
  Pt #01 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #01 Physical Functioning : Visit 10 | NA — Data not collected
  Pt #01 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #01 Role-physical : Visit 1 | 0
  Pt #01 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #01 Role-physical : Visit 5 | 25
  Pt #01 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #01 Role-physical : Visit 8 | NA — Data not collected
  Pt #01 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #01 Role-physical : Visit 9 | NA — Data not collected
  Pt #01 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #01 Role-physical : Visit 10 | NA — Data not collected
  Pt #01 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #01 Role-emotional : Visit 1 | 100
  Pt #01 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #01 Role-emotional : Visit 5 | 66.67
  Pt #01 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #01 Role-emotional : Visit 8 | NA — Data not collected
  Pt #01 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #01 Role-emotional : Visit 9 | NA — Data not collected
  Pt #01 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #01 Role-emotional : Visit 10 | NA — Data not collected
  Pt #01 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #01 Energy/fatigue : Visit 1 | 50
  Pt #01 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #01 Energy/fatigue : Visit 5 | 35
  Pt #01 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #01 Energy/fatigue : Visit 8 | NA — Data not collected
  Pt #01 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #01 Energy/fatigue : Visit 9 | NA — Data not collected
  Pt #01 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #01 Energy/fatigue : Visit 10 | NA — Data not collected
  Pt #01 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #01 Emotional Well-being : Visit 1 | 88
  Pt #01 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #01 Emotional Well-being : Visit 5 | 84
  Pt #01 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #01 Emotional Well-being : Visit 8 | NA — Data not collected
  Pt #01 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #01 Emotional Well-being : Visit 9 | NA — Data not collected
  Pt #01 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #01 Emotional Well-being : Visit 10 | NA — Data not collected
  Pt #01 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #01 Social Functioning : Visit 1 | 87.5
  Pt #01 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #01 Social Functioning : Visit 5 | 75
  Pt #01 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #01 Social Functioning : Visit 8 | NA — Data not collected
  Pt #01 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #01 Social Functioning : Visit 9 | NA — Data not collected
  Pt #01 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #01 Social Functioning : Visit 10 | NA — Data not collected
  Pt #01 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #01 Pain : Visit 1 | 100
  Pt #01 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #01 Pain : Visit 5 | 55
  Pt #01 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #01 Pain : Visit 8 | NA — Data not collected
  Pt #01 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #01 Pain : Visit 9 | NA — Data not collected
  Pt #01 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #01 Pain : Visit 10 | NA — Data not collected
  Pt #01 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #01 General Health : Visit 1 | 65
  Pt #01 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #01 General Health : Visit 5 | 55
  Pt #01 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #01 General Health : Visit 8 | NA — Data not collected
  Pt #01 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #01 General Health : Visit 9 | NA — Data not collected
  Pt #01 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #01 General Health : Visit 10 | NA — Data not collected
  Pt #2 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #2 Physical Functioning : Visit 1 | 30
  Pt #2 Physical Functioning : Visit 5 | NA — Data not collected
  Pt #2 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #2 Physical Functioning : Visit 8 | 30
  Pt #2 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #2 Physical Functioning : Visit 9 | 30
  Pt #2 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #2 Physical Functioning : Visit 10 | 75
  Pt #2 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #2 Role-physical : Visit 1 | 0
  Pt #2 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #2 Role-physical : Visit 5 | NA — Data not collected
  Pt #2 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #2 Role-physical : Visit 8 | 0
  Pt #2 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #2 Role-physical : Visit 9 | 0
  Pt #2 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #2 Role-physical : Visit 10 | 100
  Pt #2 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #2 Role-emotional : Visit 1 | 0
  Pt #2 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #2 Role-emotional : Visit 5 | NA — Data not collected
  Pt #2 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #2 Role-emotional : Visit 8 | 100
  Pt #2 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #2 Role-emotional : Visit 9 | 100
  Pt #2 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #2 Role-emotional : Visit 10 | 100
  Pt #2 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #2 Energy/fatigue : Visit 1 | 25
  Pt #2 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #2 Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #2 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #2 Energy/fatigue : Visit 8 | 40
  Pt #2 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #2 Energy/fatigue : Visit 9 | 20
  Pt #2 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #2 Energy/fatigue : Visit 10 | 55
  Pt #2 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #2 Emotional Well-being : Visit 1 | 84
  Pt #2 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #2 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #2 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #2 Emotional Well-being : Visit 8 | 88
  Pt #2 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #2 Emotional Well-being : Visit 9 | 92
  Pt #2 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #2 Emotional Well-being : Visit 10 | 76
  Pt #2 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #2 Social Functioning : Visit 1 | 87.5
  Pt #2 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #2 Social Functioning : Visit 5 | NA — Data not collected
  Pt #2 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #2 Social Functioning : Visit 8 | 87.5
  Pt #2 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #2 Social Functioning : Visit 9 | 87.5
  Pt #2 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #2 Social Functioning : Visit 10 | 87.5
  Pt #2 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #2 Pain : Visit 1 | 32.5
  Pt #2 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #2 Pain : Visit 5 | NA — Data not collected
  Pt #2 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #2 Pain : Visit 8 | 45
  Pt #2 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #2 Pain : Visit 9 | 45
  Pt #2 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #2 Pain : Visit 10 | 45
  Pt #2 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #2 General Health : Visit 1 | 25
  Pt #2 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #2 General Health : Visit 5 | NA — Data not collected
  Pt #2 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #2 General Health : Visit 8 | 35
  Pt #2 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #2 General Health : Visit 9 | 31.25
  Pt #2 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #2 General Health : Visit 10 | 30
  Pt #3 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #3 Physical Functioning : Visit 1 | 16.67
  Pt #3 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #3 Physical Functioning : Visit 5 | NA — Data not collected
  Pt #3 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #3 Physical Functioning : Visit 8 | 30
  Pt #3 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #3 Physical Functioning : Visit 9 | 40
  Pt #3 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #3 Physical Functioning : Visit 10 | 30
  Pt #3: Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #3: Role-physical : Visit 1 | 25
  Pt #3: Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #3: Role-physical : Visit 5 | NA — Data not collected
  Pt #3: Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #3: Role-physical : Visit 8 | 0
  Pt #3: Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #3: Role-physical : Visit 9 | 0
  Pt #3: Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #3: Role-physical : Visit 10 | 0
  Pt #3: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #3: Role-emotional : Visit 1 | NA — Data not collected
  Pt #3: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #3: Role-emotional : Visit 5 | NA — Data not collected
  Pt #3: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #3: Role-emotional : Visit 8 | 100
  Pt #3: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #3: Role-emotional : Visit 9 | 100
  Pt #3: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #3: Role-emotional : Visit 10 | 100
  Pt #3: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #3: Energy/fatigue : Visit 1 | 20
  Pt #3: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #3: Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #3: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #3: Energy/fatigue : Visit 8 | 5
  Pt #3: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #3: Energy/fatigue : Visit 9 | 5
  Pt #3: Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #3: Energy/fatigue : Visit 10 | 5
  Pt #3: Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #3: Emotional Well-being : Visit 1 | 88
  Pt #3: Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #3: Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #3: Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #3: Emotional Well-being : Visit 8 | 68
  Pt #3: Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #3: Emotional Well-being : Visit 9 | 68
  Pt #3: Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #3: Emotional Well-being : Visit 10 | 72
  Pt #3 : Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #3 : Social Functioning : Visit 1 | 75
  Pt #3 : Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #3 : Social Functioning : Visit 5 | NA — Data not collected
  Pt #3 : Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #3 : Social Functioning : Visit 8 | 62.5
  Pt #3 : Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #3 : Social Functioning : Visit 9 | 87.5
  Pt #3 : Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #3 : Social Functioning : Visit 10 | 75
  Pt #3 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #3 Pain : Visit 1 | 90
  Pt #3 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #3 Pain : Visit 5 | NA — Data not collected
  Pt #3 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #3 Pain : Visit 8 | 100
  Pt #3 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #3 Pain : Visit 9 | 100
  Pt #3 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #3 Pain : Visit 10 | 90
  Pt #3 : General Health : Visit 1: number analyzed (Participants) | 1
  Pt #3 : General Health : Visit 1 | 10
  Pt #3 : General Health : Visit 5: number analyzed (Participants) | 1
  Pt #3 : General Health : Visit 5 | 20
  Pt #3 : General Health : Visit 8: number analyzed (Participants) | 1
  Pt #3 : General Health : Visit 8 | 31.25
  Pt #3 : General Health : Visit 9: number analyzed (Participants) | 1
  Pt #3 : General Health : Visit 9 | 20
  Pt #3 : General Health : Visit 10: number analyzed (Participants) | 1
  Pt #3 : General Health : Visit 10 | 20
  Pt #4 : Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Physical Functioning : Visit 1 | 45
  Pt #4 : Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Physical Functioning : Visit 5 | 60
  Pt #4 : Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Physical Functioning : Visit 8 | 33.33
  Pt #4 : Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Physical Functioning : Visit 9 | 50
  Pt #4 : Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Physical Functioning : Visit 10 | 50
  Pt #4 : Role-physcial : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Role-physcial : Visit 1 | NA — Data not collected
  Pt #4 : Role-physcial : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Role-physcial : Visit 5 | 25
  Pt #4 : Role-physcial : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Role-physcial : Visit 8 | 100
  Pt #4 : Role-physcial : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Role-physcial : Visit 9 | NA — Data not collected
  Pt #4 : Role-physcial : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Role-physcial : Visit 10 | 75
  Pt #4 : Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Role-emotional : Visit 1 | 33.33
  Pt #4 : Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Role-emotional : Visit 5 | 0
  Pt #4 : Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Role-emotional : Visit 8 | 0
  Pt #4 : Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Role-emotional : Visit 9 | 33.33
  Pt #4 : Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Role-emotional : Visit 10 | 33.33
  Pt #4 : Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Energy/fatigue : Visit 1 | 25
  Pt #4 : Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Energy/fatigue : Visit 5 | 35
  Pt #4 : Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Energy/fatigue : Visit 8 | 35
  Pt #4 : Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Energy/fatigue : Visit 9 | 30
  Pt #4 : Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Energy/fatigue : Visit 10 | 35
  Pt #4 : Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Emotional Well-being : Visit 1 | 60
  Pt #4 : Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Emotional Well-being : Visit 5 | 56
  Pt #4 : Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Emotional Well-being : Visit 8 | 72
  Pt #4 : Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Emotional Well-being : Visit 9 | 66.67
  Pt #4 : Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Emotional Well-being : Visit 10 | 60
  Pt #4 : Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Social Functioning : Visit 1 | 25
  Pt #4 : Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Social Functioning : Visit 5 | 37.5
  Pt #4 : Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Social Functioning : Visit 8 | 50
  Pt #4 : Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Social Functioning : Visit 9 | NA — Data not collected
  Pt #4 : Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Social Functioning : Visit 10 | 50
  Pt #4 : Pain : Visit 1: number analyzed (Participants) | 1
  Pt #4 : Pain : Visit 1 | 22.5
  Pt #4 : Pain : Visit 5: number analyzed (Participants) | 1
  Pt #4 : Pain : Visit 5 | 20
  Pt #4 : Pain : Visit 8: number analyzed (Participants) | 1
  Pt #4 : Pain : Visit 8 | 67.5
  Pt #4 : Pain : Visit 9: number analyzed (Participants) | 1
  Pt #4 : Pain : Visit 9 | NA — Data not collected
  Pt #4 : Pain : Visit 10: number analyzed (Participants) | 1
  Pt #4 : Pain : Visit 10 | 55
  Pt #4 : General Health : Visit 1: number analyzed (Participants) | 1
  Pt #4 : General Health : Visit 1 | 35
  Pt #4 : General Health : Visit 5: number analyzed (Participants) | 1
  Pt #4 : General Health : Visit 5 | 35
  Pt #4 : General Health : Visit 8: number analyzed (Participants) | 1
  Pt #4 : General Health : Visit 8 | 30
  Pt #4 : General Health : Visit 9: number analyzed (Participants) | 1
  Pt #4 : General Health : Visit 9 | 40
  Pt #4 : General Health : Visit 10: number analyzed (Participants) | 1
  Pt #4 : General Health : Visit 10 | 30
  Pt #5: Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #5: Physical Functioning : Visit 1 | 10
  Pt #5: Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #5: Physical Functioning : Visit 5 | 20
  Pt #5: Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #5: Physical Functioning : Visit 8 | 15
  Pt #5: Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #5: Physical Functioning : Visit 9 | 10
  Pt #5: Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #5: Physical Functioning : Visit 10 | 15
  Pt #5: Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #5: Role-physical : Visit 1 | 0
  Pt #5: Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #5: Role-physical : Visit 5 | 0
  Pt #5: Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #5: Role-physical : Visit 8 | 0
  Pt #5: Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #5: Role-physical : Visit 9 | 0
  Pt #5: Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #5: Role-physical : Visit 10 | 0
  Pt #5: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #5: Role-emotional : Visit 1 | 33.33
  Pt #5: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #5: Role-emotional : Visit 5 | 0
  Pt #5: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #5: Role-emotional : Visit 8 | 33.33
  Pt #5: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #5: Role-emotional : Visit 9 | 33.33
  Pt #5: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #5: Role-emotional : Visit 10 | 33.33
  Pt #5: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #5: Energy/fatigue : Visit 1 | 25
  Pt #5: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #5: Energy/fatigue : Visit 5 | 30
  Pt #5: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #5: Energy/fatigue : Visit 8 | 20
  Pt #5: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #5: Energy/fatigue : Visit 9 | 0
  Pt #5: Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #5: Energy/fatigue : Visit 10 | 15
  Pt #5: Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #5: Emotional Well-being : Visit 1 | 72
  Pt #5: Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #5: Emotional Well-being : Visit 5 | 76
  Pt #5: Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #5: Emotional Well-being : Visit 8 | 68
  Pt #5: Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #5: Emotional Well-being : Visit 9 | 64
  Pt #5: Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #5: Emotional Well-being : Visit 10 | 68
  Pt #5: Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #5: Social Functioning : Visit 1 | 12.5
  Pt #5: Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #5: Social Functioning : Visit 5 | 50
  Pt #5: Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #5: Social Functioning : Visit 8 | 37.5
  Pt #5: Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #5: Social Functioning : Visit 9 | 12.5
  Pt #5: Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #5: Social Functioning : Visit 10 | 12.5
  Pt #5: Pain : Visit 1: number analyzed (Participants) | 1
  Pt #5: Pain : Visit 1 | 22.5
  Pt #5: Pain : Visit 5: number analyzed (Participants) | 1
  Pt #5: Pain : Visit 5 | 35
  Pt #5: Pain : Visit 8: number analyzed (Participants) | 1
  Pt #5: Pain : Visit 8 | 22.5
  Pt #5: Pain : Visit 9: number analyzed (Participants) | 1
  Pt #5: Pain : Visit 9 | 32.5
  Pt #5: Pain : Visit 10: number analyzed (Participants) | 1
  Pt #5: Pain : Visit 10 | 10
  Pt #5: General Health : Visit 1: number analyzed (Participants) | 1
  Pt #5: General Health : Visit 1 | 25
  Pt #5: General Health : Visit 5: number analyzed (Participants) | 1
  Pt #5: General Health : Visit 5 | 20
  Pt #5: General Health : Visit 8: number analyzed (Participants) | 1
  Pt #5: General Health : Visit 8 | 15
  Pt #5: General Health : Visit 9: number analyzed (Participants) | 1
  Pt #5: General Health : Visit 9 | 20
  Pt #5: General Health : Visit 10: number analyzed (Participants) | 1
  Pt #5: General Health : Visit 10 | 25
  Pt #6: Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #6: Physical Functioning : Visit 1 | 22.22
  Pt #6: Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #6: Physical Functioning : Visit 5 | 27.78
  Pt #6: Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #6: Physical Functioning : Visit 8 | 20
  Pt #6: Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #6: Physical Functioning : Visit 9 | 15
  Pt #6: Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #6: Physical Functioning : Visit 10 | 0
  Pt #6: Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #6: Role-physical : Visit 1 | NA — Data not collected
  Pt #6: Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #6: Role-physical : Visit 5 | NA — Data not collected
  Pt #6: Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #6: Role-physical : Visit 8 | 0
  Pt #6: Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #6: Role-physical : Visit 9 | 0
  Pt #6: Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #6: Role-physical : Visit 10 | 0
  Pt #6: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #6: Role-emotional : Visit 1 | NA — Data not collected
  Pt #6: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #6: Role-emotional : Visit 5 | NA — Data not collected
  Pt #6: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #6: Role-emotional : Visit 8 | 0
  Pt #6: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #6: Role-emotional : Visit 9 | 100
  Pt #6: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #6: Role-emotional : Visit 10 | 33.3
  Pt #6: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #6: Energy/fatigue : Visit 1 | 10
  Pt #6: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #6: Energy/fatigue : Visit 5 | 10
  Pt #6: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #6: Energy/fatigue : Visit 8 | 15
  Pt #6: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #6: Energy/fatigue : Visit 9 | 10
  Pt #6: Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #6: Energy/fatigue : Visit 10 | 0
  Pt #6: Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #6: Emotional Well-being : Visit 1 | 46.67
  Pt #6: Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #6: Emotional Well-being : Visit 5 | 60
  Pt #6: Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #6: Emotional Well-being : Visit 8 | 64
  Pt #6: Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #6: Emotional Well-being : Visit 9 | 64
  Pt #6: Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #6: Emotional Well-being : Visit 10 | 36
  Pt #6: Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #6: Social Functioning : Visit 1 | NA — Data not collected
  Pt #6: Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #6: Social Functioning : Visit 5 | NA — Data not collected
  Pt #6: Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #6: Social Functioning : Visit 8 | 25
  Pt #6: Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #6: Social Functioning : Visit 9 | 37.5
  Pt #6: Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #6: Social Functioning : Visit 10 | 25
  Pt #6: Pain : Visit 1: number analyzed (Participants) | 1
  Pt #6: Pain : Visit 1 | NA — Data not collected
  Pt #6: Pain : Visit 5: number analyzed (Participants) | 1
  Pt #6: Pain : Visit 5 | NA — Data not collected
  Pt #6: Pain : Visit 8: number analyzed (Participants) | 1
  Pt #6: Pain : Visit 8 | 100
  Pt #6: Pain : Visit 9: number analyzed (Participants) | 1
  Pt #6: Pain : Visit 9 | 100
  Pt #6: Pain : Visit 10: number analyzed (Participants) | 1
  Pt #6: Pain : Visit 10 | 55
  Pt #6: General Health : Visit 1: number analyzed (Participants) | 1
  Pt #6: General Health : Visit 1 | 20
  Pt #6: General Health : Visit 5: number analyzed (Participants) | 1
  Pt #6: General Health : Visit 5 | 20
  Pt #6: General Health : Visit 8: number analyzed (Participants) | 1
  Pt #6: General Health : Visit 8 | 20
  Pt #6: General Health : Visit 9: number analyzed (Participants) | 1
  Pt #6: General Health : Visit 9 | 15
  Pt #6: General Health : Visit 10: number analyzed (Participants) | 1
  Pt #6: General Health : Visit 10 | 15
  Pt #7: Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #7: Physical Functioning : Visit 1 | 20
  Pt #7: Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #7: Physical Functioning : Visit 5 | 55
  Pt #7: Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #7: Physical Functioning : Visit 8 | NA — Data not collected
  Pt #7: Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #7: Physical Functioning : Visit 9 | NA — Data not collected
  Pt #7: Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #7: Physical Functioning : Visit 10 | NA — Data not collected
  Pt #7: Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #7: Role-physical : Visit 1 | 100
  Pt #7: Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #7: Role-physical : Visit 5 | 25
  Pt #7: Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #7: Role-physical : Visit 8 | NA — Data not collected
  Pt #7: Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #7: Role-physical : Visit 9 | NA — Data not collected
  Pt #7: Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #7: Role-physical : Visit 10 | NA — Data not collected
  Pt #7: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #7: Role-emotional : Visit 1 | 100
  Pt #7: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #7: Role-emotional : Visit 5 | 100
  Pt #7: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #7: Role-emotional : Visit 8 | NA — Data not collected
  Pt #7: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #7: Role-emotional : Visit 9 | NA — Data not collected
  Pt #7: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #7: Role-emotional : Visit 10 | NA — Data not collected
  Pt #7: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #7: Energy/fatigue : Visit 1 | 65
  Pt #7: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #7: Energy/fatigue : Visit 5 | 10
  Pt #7: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #7: Energy/fatigue : Visit 8 | NA — Data not collected
  Pt #7: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #7: Energy/fatigue : Visit 9 | NA — Data not collected
  Pt #7: Energy/fatigue : Visit 10 | NA — Data not collected
  Pt #7: Emotional Well-being : Visit 1 | 72
  Pt #7: Emotional Well-being : Visit 5 | 88
  Pt #7: Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #7: Emotional Well-being : Visit 8 | NA — Data not collected
  Pt #7: Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #7: Emotional Well-being : Visit 9 | NA — Data not collected
  Pt #7: Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #7: Emotional Well-being : Visit 10 | NA — Data not collected
  Pt #7: Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #7: Social Functioning : Visit 1 | 50
  Pt #7: Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #7: Social Functioning : Visit 5 | 87.5
  Pt #7: Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #7: Social Functioning : Visit 8 | NA — Data not collected
  Pt #7: Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #7: Social Functioning : Visit 9 | NA — Data not collected
  Pt #7: Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #7: Social Functioning : Visit 10 | NA — Data not collected
  Pt #7: Pain : Visit 1: number analyzed (Participants) | 1
  Pt #7: Pain : Visit 1 | 77.5
  Pt #7: Pain : Visit 5: number analyzed (Participants) | 1
  Pt #7: Pain : Visit 5 | 77.5
  Pt #7: Pain : Visit 8: number analyzed (Participants) | 1
  Pt #7: Pain : Visit 8 | NA — Data not collected
  Pt #7: Pain : Visit 9: number analyzed (Participants) | 1
  Pt #7: Pain : Visit 9 | NA — Data not collected
  Pt #7: Pain : Visit 10: number analyzed (Participants) | 1
  Pt #7: Pain : Visit 10 | NA — Data not collected
  Pt #7: General Health : Visit 1: number analyzed (Participants) | 1
  Pt #7: General Health : Visit 1 | 30
  Pt #7: General Health : Visit 5: number analyzed (Participants) | 1
  Pt #7: General Health : Visit 5 | 35
  Pt #7: General Health : Visit 8: number analyzed (Participants) | 1
  Pt #7: General Health : Visit 8 | NA — Data not collected
  Pt #7: General Health : Visit 9: number analyzed (Participants) | 1
  Pt #7: General Health : Visit 9 | NA — Data not collected
  Pt #7: General Health : Visit 10: number analyzed (Participants) | 1
  Pt #7: General Health : Visit 10 | NA — Data not collected
  Pt #8: Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #8: Physical Functioning : Visit 1 | 45
  Pt #8: Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #8: Physical Functioning : Visit 5 | 75
  Pt #8: Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #8: Physical Functioning : Visit 8 | 45
  Pt #8: Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #8: Physical Functioning : Visit 9 | 70
  Pt #8: Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #8: Physical Functioning : Visit 10 | 45
  Pt #8 Role-physcial : Visit 1: number analyzed (Participants) | 1
  Pt #8 Role-physcial : Visit 1 | 0
  Pt #8 Role-physcial : Visit 5: number analyzed (Participants) | 1
  Pt #8 Role-physcial : Visit 5 | 33.33
  Pt #8 Role-physcial : Visit 8: number analyzed (Participants) | 1
  Pt #8 Role-physcial : Visit 8 | 66.67
  Pt #8 Role-physcial : Visit 9: number analyzed (Participants) | 1
  Pt #8 Role-physcial : Visit 9 | 100
  Pt #8 Role-physcial : Visit 10: number analyzed (Participants) | 1
  Pt #8 Role-physcial : Visit 10 | 100
  Pt #8: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #8: Role-emotional : Visit 1 | 0
  Pt #8: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #8: Role-emotional : Visit 5 | 50
  Pt #8: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #8: Role-emotional : Visit 8 | 50
  Pt #8: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #8: Role-emotional : Visit 9 | 45
  Pt #8: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #8: Role-emotional : Visit 10 | 50
  Pt #8: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #8: Energy/fatigue : Visit 1 | 40
  Pt #8: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #8: Energy/fatigue : Visit 5 | 50
  Pt #8: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #8: Energy/fatigue : Visit 8 | 50
  Pt #8: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #8: Energy/fatigue : Visit 9 | 45
  Pt #8: Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #8: Energy/fatigue : Visit 10 | 50
  Pt #8 : Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #8 : Emotional Well-being : Visit 1 | 52
  Pt #8 : Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #8 : Emotional Well-being : Visit 5 | 60
  Pt #8 : Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #8 : Emotional Well-being : Visit 8 | 52
  Pt #8 : Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #8 : Emotional Well-being : Visit 9 | 92
  Pt #8 : Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #8 : Emotional Well-being : Visit 10 | 92
  Pt #8: Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #8: Social Functioning : Visit 1 | 50
  Pt #8: Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #8: Social Functioning : Visit 5 | 50
  Pt #8: Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #8: Social Functioning : Visit 8 | 50
  Pt #8: Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #8: Social Functioning : Visit 9 | 75
  Pt #8: Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #8: Social Functioning : Visit 10 | 87.5
  Pt #8 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #8 Pain : Visit 1 | 45
  Pt #8 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #8 Pain : Visit 5 | 45
  Pt #8 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #8 Pain : Visit 8 | 45
  Pt #8 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #8 Pain : Visit 9 | 80
  Pt #8 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #8 Pain : Visit 10 | 90
  Pt #8: General Health : Visit 1: number analyzed (Participants) | 1
  Pt #8: General Health : Visit 1 | 45
  Pt #8: General Health : Visit 5: number analyzed (Participants) | 1
  Pt #8: General Health : Visit 5 | 50
  Pt #8: General Health : Visit 8: number analyzed (Participants) | 1
  Pt #8: General Health : Visit 8 | 55
  Pt #8: General Health : Visit 9: number analyzed (Participants) | 1
  Pt #8: General Health : Visit 9 | 80
  Pt #8: General Health : Visit 10: number analyzed (Participants) | 1
  Pt #8: General Health : Visit 10 | 65
  Pt #9: Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #9: Physical Functioning : Visit 1 | 75
  Pt #9: Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #9: Physical Functioning : Visit 5 | NA — Data not collected
  Pt #9: Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #9: Physical Functioning : Visit 8 | 70
  Pt #9: Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #9: Physical Functioning : Visit 9 | 70
  Pt #9: Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #9: Physical Functioning : Visit 10 | 80
  Pt #9: Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #9: Role-physical : Visit 1 | 0
  Pt #9: Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #9: Role-physical : Visit 5 | NA — Data not collected
  Pt #9: Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #9: Role-physical : Visit 8 | 0
  Pt #9: Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #9: Role-physical : Visit 9 | 25
  Pt #9: Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #9: Role-physical : Visit 10 | 100
  Pt #9: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #9: Role-emotional : Visit 1 | 100
  Pt #9: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #9: Role-emotional : Visit 5 | NA — Data not collected
  Pt #9: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #9: Role-emotional : Visit 8 | 100
  Pt #9: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #9: Role-emotional : Visit 9 | 100
  Pt #9: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #9: Role-emotional : Visit 10 | 100
  Pt #9: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #9: Energy/fatigue : Visit 1 | 70
  Pt #9: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #9: Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #9: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #9: Energy/fatigue : Visit 8 | 60
  Pt #9: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #9: Energy/fatigue : Visit 9 | 70
  Pt #9: Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #9: Energy/fatigue : Visit 10 | 75
  Pt #9: Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #9: Emotional Well-being : Visit 1 | 84
  Pt #9: Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #9: Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #9: Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #9: Emotional Well-being : Visit 8 | 80
  Pt #9: Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #9: Emotional Well-being : Visit 9 | 92
  Pt #9: Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #9: Emotional Well-being : Visit 10 | 80
  Pt #9: Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #9: Social Functioning : Visit 1 | 75
  Pt #9: Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #9: Social Functioning : Visit 5 | NA — Data not collected
  Pt #9: Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #9: Social Functioning : Visit 8 | 62.5
  Pt #9: Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #9: Social Functioning : Visit 9 | 87.5
  Pt #9: Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #9: Social Functioning : Visit 10 | 75
  Pt #9: Pain : Visit 1: number analyzed (Participants) | 1
  Pt #9: Pain : Visit 1 | 77.5
  Pt #9: Pain : Visit 5: number analyzed (Participants) | 1
  Pt #9: Pain : Visit 5 | NA — Data not collected
  Pt #9: Pain : Visit 8: number analyzed (Participants) | 1
  Pt #9: Pain : Visit 8 | 45
  Pt #9: Pain : Visit 9: number analyzed (Participants) | 1
  Pt #9: Pain : Visit 9 | 77.5
  Pt #9: Pain : Visit 10: number analyzed (Participants) | 1
  Pt #9: Pain : Visit 10 | 67.5
  Pt #9: General Health : Visit 1: number analyzed (Participants) | 1
  Pt #9: General Health : Visit 1 | 70
  Pt #9: General Health : Visit 5: number analyzed (Participants) | 1
  Pt #9: General Health : Visit 5 | NA — Data not collected
  Pt #9: General Health : Visit 8: number analyzed (Participants) | 1
  Pt #9: General Health : Visit 8 | 31.25
  Pt #9: General Health : Visit 9: number analyzed (Participants) | 1
  Pt #9: General Health : Visit 9 | 40
  Pt #9: General Health : Visit 10: number analyzed (Participants) | 1
  Pt #9: General Health : Visit 10 | 56.25
  Pt #10: Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #10: Physical Functioning : Visit 1 | 80
  Pt #10: Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #10: Physical Functioning : Visit 5 | 90
  Pt #10: Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #10: Physical Functioning : Visit 8 | 83.33
  Pt #10: Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #10: Physical Functioning : Visit 9 | 85
  Pt #10: Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #10: Physical Functioning : Visit 10 | 85
  Pt #10: Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #10: Role-physical : Visit 1 | 0
  Pt #10: Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #10: Role-physical : Visit 5 | 25
  Pt #10: Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #10: Role-physical : Visit 8 | 100
  Pt #10: Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #10: Role-physical : Visit 9 | 25
  Pt #10: Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #10: Role-physical : Visit 10 | 100
  Pt #10: Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #10: Role-emotional : Visit 1 | 100
  Pt #10: Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #10: Role-emotional : Visit 5 | 100
  Pt #10: Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #10: Role-emotional : Visit 8 | 100
  Pt #10: Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #10: Role-emotional : Visit 9 | 100
  Pt #10: Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #10: Role-emotional : Visit 10 | 100
  Pt #10: Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #10: Energy/fatigue : Visit 1 | 60
  Pt #10: Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #10: Energy/fatigue : Visit 5 | 75
  Pt #10: Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #10: Energy/fatigue : Visit 8 | 80
  Pt #10: Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #10: Energy/fatigue : Visit 9 | 65
  Pt #10: Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #10: Energy/fatigue : Visit 10 | 80
  Pt #10: Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #10: Emotional Well-being : Visit 1 | 88
  Pt #10: Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #10: Emotional Well-being : Visit 5 | 84
  Pt #10: Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #10: Emotional Well-being : Visit 8 | 84
  Pt #10: Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #10: Emotional Well-being : Visit 9 | 92
  Pt #10: Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #10: Emotional Well-being : Visit 10 | 92
  Pt #10 : Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #10 : Social Functioning : Visit 1 | 87.5
  Pt #10 : Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #10 : Social Functioning : Visit 5 | 87.5
  Pt #10 : Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #10 : Social Functioning : Visit 8 | 87.5
  Pt #10 : Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #10 : Social Functioning : Visit 9 | 75
  Pt #10 : Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #10 : Social Functioning : Visit 10 | 87.5
  Pt #10 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #10 Pain : Visit 1 | 100
  Pt #10 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #10 Pain : Visit 5 | 77.5
  Pt #10 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #10 Pain : Visit 8 | 77.5
  Pt #10 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #10 Pain : Visit 9 | 77.5
  Pt #10 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #10 Pain : Visit 10 | 100
  Pt #10 Visit 1 : General Health : Visit 1: number analyzed (Participants) | 1
  Pt #10 Visit 1 : General Health : Visit 1 | 80
  Pt #10 Visit 1 : General Health : Visit 5: number analyzed (Participants) | 1
  Pt #10 Visit 1 : General Health : Visit 5 | 65
  Pt #10 Visit 1 : General Health : Visit 8: number analyzed (Participants) | 1
  Pt #10 Visit 1 : General Health : Visit 8 | 65
  Pt #10 Visit 1 : General Health : Visit 9: number analyzed (Participants) | 1
  Pt #10 Visit 1 : General Health : Visit 9 | 65
  Pt #10 Visit 1 : General Health : Visit 10: number analyzed (Participants) | 1
  Pt #10 Visit 1 : General Health : Visit 10 | 65
  Pt #11 Visit 1 : Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Physical Functioning : Visit 1 | 15
  Pt #11 Visit 1 : Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Physical Functioning : Visit 5 | NA — Data not collected
  Pt #11 Visit 1 : Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Physical Functioning : Visit 8 | 10
  Pt #11 Visit 1 : Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Physical Functioning : Visit 9 | 5
  Pt #11 Visit 1 : Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Physical Functioning : Visit 10 | 10
  Pt #11 Visit 1 : Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-physical : Visit 1 | 25
  Pt #11 Visit 1 : Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-physical : Visit 5 | NA — Data not collected
  Pt #11 Visit 1 : Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-physical : Visit 8 | 25
  Pt #11 Visit 1 : Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-physical : Visit 9 | 0
  Pt #11 Visit 1 : Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-physical : Visit 10 | 25
  Pt #11 Visit 1 : Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-emotional : Visit 1 | 0
  Pt #11 Visit 1 : Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-emotional : Visit 5 | NA — Data not collected
  Pt #11 Visit 1 : Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-emotional : Visit 8 | 100
  Pt #11 Visit 1 : Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-emotional : Visit 9 | 0
  Pt #11 Visit 1 : Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Role-emotional : Visit 10 | 66.67
  Pt #11 Visit 1 : Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Energy/fatigue : Visit 1 | 30
  Pt #11 Visit 1 : Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #11 Visit 1 : Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Energy/fatigue : Visit 8 | 40
  Pt #11 Visit 1 : Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Energy/fatigue : Visit 9 | 20
  Pt #11 Visit 1 : Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Energy/fatigue : Visit 10 | 20
  Pt #11 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #11 Emotional Well-being : Visit 1 | 60
  Pt #11 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #11 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #11 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #11 Emotional Well-being : Visit 8 | 84
  Pt #11 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #11 Emotional Well-being : Visit 9 | 60
  Pt #11 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #11 Emotional Well-being : Visit 10 | 68
  Pt #11 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #11 Social Functioning : Visit 1 | 50
  Pt #11 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #11 Social Functioning : Visit 5 | NA — Data not collected
  Pt #11 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #11 Social Functioning : Visit 8 | 87.5
  Pt #11 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #11 Social Functioning : Visit 9 | 37.5
  Pt #11 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #11 Social Functioning : Visit 10 | 62.5
  Pt #11 Visit 1 : Pain : Visit 1: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Pain : Visit 1 | 0
  Pt #11 Visit 1 : Pain : Visit 5: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Pain : Visit 5 | NA — Data not collected
  Pt #11 Visit 1 : Pain : Visit 8: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Pain : Visit 8 | 22.5
  Pt #11 Visit 1 : Pain : Visit 9: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Pain : Visit 9 | 10
  Pt #11 Visit 1 : Pain : Visit 10: number analyzed (Participants) | 1
  Pt #11 Visit 1 : Pain : Visit 10 | 22.5
  Pt #11 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #11 General Health : Visit 1 | 5
  Pt #11 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #11 General Health : Visit 5 | NA — Data not collected
  Pt #11 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #11 General Health : Visit 8 | 15
  Pt #11 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #11 General Health : Visit 9 | 10
  Pt #11 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #11 General Health : Visit 10 | 15
  Pt #12 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #12 Physical Functioning : Visit 1 | 35
  Pt #12 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #12 Physical Functioning : Visit 5 | 50
  Pt #12 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #12 Physical Functioning : Visit 8 | NA — Data not collected
  Pt #12 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #12 Physical Functioning : Visit 9 | 40
  Pt #12 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #12 Physical Functioning : Visit 10 | 44.44
  Pt #12 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #12 Role-physical : Visit 1 | 0
  Pt #12 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #12 Role-physical : Visit 5 | 0
  Pt #12 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #12 Role-physical : Visit 8 | NA — Data not collected
  Pt #12 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #12 Role-physical : Visit 9 | 75
  Pt #12 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #12 Role-physical : Visit 10 | 0
  Pt #12 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #12 Role-emotional : Visit 1 | 33.33
  Pt #12 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #12 Role-emotional : Visit 5 | 100
  Pt #12 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #12 Role-emotional : Visit 8 | NA — Data not collected
  Pt #12 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #12 Role-emotional : Visit 9 | 100
  Pt #12 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #12 Role-emotional : Visit 10 | 100
  Pt #12 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #12 Energy/fatigue : Visit 1 | 40
  Pt #12 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #12 Energy/fatigue : Visit 5 | 60
  Pt #12 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #12 Energy/fatigue : Visit 8 | NA — Data not collected
  Pt #12 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #12 Energy/fatigue : Visit 9 | 65
  Pt #12 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #12 Energy/fatigue : Visit 10 | 70
  Pt #12 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #12 Emotional Well-being : Visit 1 | 68
  Pt #12 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #12 Emotional Well-being : Visit 5 | 80
  Pt #12 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #12 Emotional Well-being : Visit 8 | NA — Data not collected
  Pt #12 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #12 Emotional Well-being : Visit 9 | 72
  Pt #12 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #12 Emotional Well-being : Visit 10 | 80
  Pt #12 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #12 Social Functioning : Visit 1 | 50
  Pt #12 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #12 Social Functioning : Visit 5 | 87.5
  Pt #12 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #12 Social Functioning : Visit 8 | NA — Data not collected
  Pt #12 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #12 Social Functioning : Visit 9 | 87.5
  Pt #12 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #12 Social Functioning : Visit 10 | 87.5
  Pt #12 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #12 Pain : Visit 1 | 77.5
  Pt #12 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #12 Pain : Visit 5 | 55
  Pt #12 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #12 Pain : Visit 8 | NA — Data not collected
  Pt #12 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #12 Pain : Visit 9 | 67.5
  Pt #12 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #12 Pain : Visit 10 | 77.5
  Pt #12 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #12 General Health : Visit 1 | 60
  Pt #12 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #12 General Health : Visit 5 | 45
  Pt #12 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #12 General Health : Visit 8 | NA — Data not collected
  Pt #12 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #12 General Health : Visit 9 | 50
  Pt #12 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #12 General Health : Visit 10 | 55
  Pt#13 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt#13 Physical Functioning : Visit 1 | 20
  Pt#13 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt#13 Physical Functioning : Visit 5 | NA — Data not collected
  Pt#13 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt#13 Physical Functioning : Visit 8 | 15
  Pt#13 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt#13 Physical Functioning : Visit 9 | 10
  Pt#13 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt#13 Physical Functioning : Visit 10 | 15
  Pt #13 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #13 Role-physical : Visit 1 | 25
  Pt #13 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #13 Role-physical : Visit 5 | NA — Data not collected
  Pt #13 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #13 Role-physical : Visit 8 | 0
  Pt #13 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #13 Role-physical : Visit 9 | 0
  Pt #13 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #13 Role-physical : Visit 10 | 0
  Pt #13 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #13 Role-emotional : Visit 1 | 33.33
  Pt #13 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #13 Role-emotional : Visit 5 | NA — Data not collected
  Pt #13 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #13 Role-emotional : Visit 8 | 0
  Pt #13 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #13 Role-emotional : Visit 9 | 100
  Pt #13 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #13 Role-emotional : Visit 10 | 100
  Pt #13 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #13 Energy/fatigue : Visit 1 | 40
  Pt #13 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #13 Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #13 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #13 Energy/fatigue : Visit 8 | 25
  Pt #13 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #13 Energy/fatigue : Visit 9 | 25
  Pt #13 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #13 Energy/fatigue : Visit 10 | 10
  Pt #13 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #13 Emotional Well-being : Visit 1 | 60
  Pt #13 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #13 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #13 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #13 Emotional Well-being : Visit 8 | 60
  Pt #13 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #13 Emotional Well-being : Visit 9 | 64
  Pt #13 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #13 Emotional Well-being : Visit 10 | 72
  Pt #13 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #13 Social Functioning : Visit 1 | 62.5
  Pt #13 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #13 Social Functioning : Visit 5 | NA — Data not collected
  Pt #13 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #13 Social Functioning : Visit 8 | 62.5
  Pt #13 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #13 Social Functioning : Visit 9 | 62.5
  Pt #13 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #13 Social Functioning : Visit 10 | 62.5
  Pt #13 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #13 Pain : Visit 1 | 67.5
  Pt #13 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #13 Pain : Visit 5 | NA — Data not collected
  Pt #13 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #13 Pain : Visit 8 | 10
  Pt #13 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #13 Pain : Visit 9 | 32.5
  Pt #13 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #13 Pain : Visit 10 | 45
  Pt #13 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #13 General Health : Visit 1 | 20
  Pt #13 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #13 General Health : Visit 5 | NA — Data not collected
  Pt #13 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #13 General Health : Visit 8 | 10
  Pt #13 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #13 General Health : Visit 9 | 15
  Pt #13 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #13 General Health : Visit 10 | 15
  Pt #14 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #14 Physical Functioning : Visit 1 | 80
  Pt #14 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #14 Physical Functioning : Visit 5 | NA — Data not collected
  Pt #14 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #14 Physical Functioning : Visit 8 | 45
  Pt #14 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #14 Physical Functioning : Visit 9 | 50
  Pt #14 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #14 Physical Functioning : Visit 10 | 60
  Pt #14 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #14 Role-physical : Visit 1 | 100
  Pt #14 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #14 Role-physical : Visit 5 | NA — Data not collected
  Pt #14 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #14 Role-physical : Visit 8 | 0
  Pt #14 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #14 Role-physical : Visit 9 | 0
  Pt #14 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #14 Role-physical : Visit 10 | 50
  Pt #14 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #14 Role-emotional : Visit 1 | 0
  Pt #14 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #14 Role-emotional : Visit 5 | NA — Data not collected
  Pt #14 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #14 Role-emotional : Visit 8 | 0
  Pt #14 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #14 Role-emotional : Visit 9 | 33.33
  Pt #14 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #14 Role-emotional : Visit 10 | 100
  Pt #14 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #14 Energy/fatigue : Visit 1 | 60
  Pt #14 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #14 Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #14 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #14 Energy/fatigue : Visit 8 | 50
  Pt #14 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #14 Energy/fatigue : Visit 9 | 35
  Pt #14 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #14 Energy/fatigue : Visit 10 | 75
  Pt #14 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #14 Emotional Well-being : Visit 1 | 56
  Pt #14 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #14 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #14 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #14 Emotional Well-being : Visit 8 | 64
  Pt #14 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #14 Emotional Well-being : Visit 9 | 52
  Pt #14 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #14 Emotional Well-being : Visit 10 | 92
  Pt #14 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #14 Social Functioning : Visit 1 | 100
  Pt #14 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #14 Social Functioning : Visit 5 | NA — Data not collected
  Pt #14 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #14 Social Functioning : Visit 8 | 62.5
  Pt #14 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #14 Social Functioning : Visit 9 | 62.5
  Pt #14 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #14 Social Functioning : Visit 10 | 62.5
  Pt #14 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #14 Pain : Visit 1 | 100
  Pt #14 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #14 Pain : Visit 5 | NA — Data not collected
  Pt #14 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #14 Pain : Visit 8 | 32.5
  Pt #14 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #14 Pain : Visit 9 | 45
  Pt #14 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #14 Pain : Visit 10 | 32.5
  Pt #14 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #14 General Health : Visit 1 | 50
  Pt #14 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #14 General Health : Visit 5 | NA — Data not collected
  Pt #14 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #14 General Health : Visit 8 | 50
  Pt #14 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #14 General Health : Visit 9 | 40
  Pt #14 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #14 General Health : Visit 10 | 60
  Pt #15 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #15 Physical Functioning : Visit 1 | 10
  Pt #15 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #15 Physical Functioning : Visit 5 | NA — Data not collected
  Pt #15 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #15 Physical Functioning : Visit 8 | NA — Data not collected
  Pt #15 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #15 Physical Functioning : Visit 9 | 5
  Pt #15 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #15 Physical Functioning : Visit 10 | 11.11
  Pt #15 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #15 Role-physical : Visit 1 | 0
  Pt #15 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #15 Role-physical : Visit 5 | NA — Data not collected
  Pt #15 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #15 Role-physical : Visit 8 | NA — Data not collected
  Pt #15 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #15 Role-physical : Visit 9 | 0
  Pt #15 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #15 Role-physical : Visit 10 | 25
  Pt #15 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #15 Role-emotional : Visit 1 | 66.67
  Pt #15 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #15 Role-emotional : Visit 5 | NA — Data not collected
  Pt #15 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #15 Role-emotional : Visit 8 | NA — Data not collected
  Pt #15 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #15 Role-emotional : Visit 9 | 66.67
  Pt #15 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #15 Role-emotional : Visit 10 | 100
  Pt #15 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #15 Energy/fatigue : Visit 1 | 0
  Pt #15 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #15 Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #15 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #15 Energy/fatigue : Visit 8 | NA — Data not collected
  Pt #15 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #15 Energy/fatigue : Visit 9 | 0
  Pt #15 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #15 Energy/fatigue : Visit 10 | 0
  Pt #15 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #15 Emotional Well-being : Visit 1 | 88
  Pt #15 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #15 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #15 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #15 Emotional Well-being : Visit 8 | NA — Data not collected
  Pt #15 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #15 Emotional Well-being : Visit 9 | 88
  Pt #15 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #15 Emotional Well-being : Visit 10 | 80
  Pt #15 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #15 Social Functioning : Visit 1 | 37.5
  Pt #15 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #15 Social Functioning : Visit 5 | NA — Data not collected
  Pt #15 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #15 Social Functioning : Visit 8 | NA — Data not collected
  Pt #15 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #15 Social Functioning : Visit 9 | 50
  Pt #15 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #15 Social Functioning : Visit 10 | 50
  Pt #15 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #15 Pain : Visit 1 | NA — Data not collected
  Pt #15 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #15 Pain : Visit 5 | NA — Data not collected
  Pt #15 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #15 Pain : Visit 8 | NA — Data not collected
  Pt #15 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #15 Pain : Visit 9 | 70
  Pt #15 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #15 Pain : Visit 10 | 22.5
  Pt #15 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #15 General Health : Visit 1 | 15
  Pt #15 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #15 General Health : Visit 5 | NA — Data not collected
  Pt #15 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #15 General Health : Visit 8 | NA — Data not collected
  Pt #15 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #15 General Health : Visit 9 | 15
  Pt #15 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #15 General Health : Visit 10 | 10
  Pt #16 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #16 Physical Functioning : Visit 1 | 30
  Pt #16 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #16 Physical Functioning : Visit 5 | NA — Data not collected
  Pt #16 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #16 Physical Functioning : Visit 8 | NA — Data not collected
  Pt #16 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #16 Physical Functioning : Visit 9 | NA — Data not collected
  Pt #16 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #16 Physical Functioning : Visit 10 | NA — Data not collected
  Pt #16 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #16 Role-physical : Visit 1 | 25
  Pt #16 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #16 Role-physical : Visit 5 | NA — Data not collected
  Pt #16 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #16 Role-physical : Visit 8 | NA — Data not collected
  Pt #16 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #16 Role-physical : Visit 9 | NA — Data not collected
  Pt #16 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #16 Role-physical : Visit 10 | NA — Data not collected
  Pt #16 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #16 Role-emotional : Visit 1 | 0
  Pt #16 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #16 Role-emotional : Visit 5 | NA — Data not collected
  Pt #16 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #16 Role-emotional : Visit 8 | NA — Data not collected
  Pt #16 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #16 Role-emotional : Visit 9 | NA — Data not collected
  Pt #16 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #16 Role-emotional : Visit 10 | NA — Data not collected
  Pt #16 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #16 Energy/fatigue : Visit 1 | 20
  Pt #16 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #16 Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #16 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #16 Energy/fatigue : Visit 8 | NA — Data not collected
  Pt #16 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #16 Energy/fatigue : Visit 9 | NA — Data not collected
  Pt #16 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #16 Energy/fatigue : Visit 10 | NA — Data not collected
  Pt #16 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #16 Emotional Well-being : Visit 1 | 48
  Pt #16 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #16 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #16 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #16 Emotional Well-being : Visit 8 | NA — Data not collected
  Pt #16 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #16 Emotional Well-being : Visit 9 | NA — Data not collected
  Pt #16 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #16 Emotional Well-being : Visit 10 | NA — Data not collected
  Pt #16 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #16 Social Functioning : Visit 1 | 0
  Pt #16 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #16 Social Functioning : Visit 5 | NA — Data not collected
  Pt #16 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #16 Social Functioning : Visit 8 | NA — Data not collected
  Pt #16 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #16 Social Functioning : Visit 9 | NA — Data not collected
  Pt #16 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #16 Social Functioning : Visit 10 | NA — Data not collected
  Pt #16 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #16 Pain : Visit 1 | 22.5
  Pt #16 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #16 Pain : Visit 5 | NA — Data not collected
  Pt #16 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #16 Pain : Visit 8 | NA — Data not collected
  Pt #16 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #16 Pain : Visit 9 | NA — Data not collected
  Pt #16 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #16 Pain : Visit 10 | NA — Data not collected
  Pt #16 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #16 General Health : Visit 1 | 25
  Pt #16 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #16 General Health : Visit 5 | NA — Data not collected
  Pt #16 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #16 General Health : Visit 8 | NA — Data not collected
  Pt #16 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #16 General Health : Visit 9 | NA — Data not collected
  Pt #16 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #16 General Health : Visit 10 | NA — Data not collected
  Pt #17 Physical Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #17 Physical Functioning : Visit 1 | 95
  Pt #17 Physical Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #17 Physical Functioning : Visit 5 | NA — Data not collected
  Pt #17 Physical Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #17 Physical Functioning : Visit 8 | 88.89
  Pt #17 Physical Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #17 Physical Functioning : Visit 9 | 85
  Pt #17 Physical Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #17 Physical Functioning : Visit 10 | NA — Data not collected
  Pt #17 Role-physical : Visit 1: number analyzed (Participants) | 1
  Pt #17 Role-physical : Visit 1 | 50
  Pt #17 Role-physical : Visit 5: number analyzed (Participants) | 1
  Pt #17 Role-physical : Visit 5 | NA — Data not collected
  Pt #17 Role-physical : Visit 8: number analyzed (Participants) | 1
  Pt #17 Role-physical : Visit 8 | 100
  Pt #17 Role-physical : Visit 9: number analyzed (Participants) | 1
  Pt #17 Role-physical : Visit 9 | 75
  Pt #17 Role-physical : Visit 10: number analyzed (Participants) | 1
  Pt #17 Role-physical : Visit 10 | NA — Data not collected
  Pt #17 Role-emotional : Visit 1: number analyzed (Participants) | 1
  Pt #17 Role-emotional : Visit 1 | 66.67
  Pt #17 Role-emotional : Visit 5: number analyzed (Participants) | 1
  Pt #17 Role-emotional : Visit 5 | NA — Data not collected
  Pt #17 Role-emotional : Visit 8: number analyzed (Participants) | 1
  Pt #17 Role-emotional : Visit 8 | 100
  Pt #17 Role-emotional : Visit 9: number analyzed (Participants) | 1
  Pt #17 Role-emotional : Visit 9 | 100
  Pt #17 Role-emotional : Visit 10: number analyzed (Participants) | 1
  Pt #17 Role-emotional : Visit 10 | NA — Data not collected
  Pt #17 Energy/fatigue : Visit 1: number analyzed (Participants) | 1
  Pt #17 Energy/fatigue : Visit 1 | 70
  Pt #17 Energy/fatigue : Visit 5: number analyzed (Participants) | 1
  Pt #17 Energy/fatigue : Visit 5 | NA — Data not collected
  Pt #17 Energy/fatigue : Visit 8: number analyzed (Participants) | 1
  Pt #17 Energy/fatigue : Visit 8 | 40
  Pt #17 Energy/fatigue : Visit 9: number analyzed (Participants) | 1
  Pt #17 Energy/fatigue : Visit 9 | 35
  Pt #17 Energy/fatigue : Visit 10: number analyzed (Participants) | 1
  Pt #17 Energy/fatigue : Visit 10 | NA — Data not collected
  Pt #17 Emotional Well-being : Visit 1: number analyzed (Participants) | 1
  Pt #17 Emotional Well-being : Visit 1 | 96
  Pt #17 Emotional Well-being : Visit 5: number analyzed (Participants) | 1
  Pt #17 Emotional Well-being : Visit 5 | NA — Data not collected
  Pt #17 Emotional Well-being : Visit 8: number analyzed (Participants) | 1
  Pt #17 Emotional Well-being : Visit 8 | 76
  Pt #17 Emotional Well-being : Visit 9: number analyzed (Participants) | 1
  Pt #17 Emotional Well-being : Visit 9 | 76
  Pt #17 Emotional Well-being : Visit 10: number analyzed (Participants) | 1
  Pt #17 Emotional Well-being : Visit 10 | NA — Data not collected
  Pt #17 Social Functioning : Visit 1: number analyzed (Participants) | 1
  Pt #17 Social Functioning : Visit 1 | 87.5
  Pt #17 Social Functioning : Visit 5: number analyzed (Participants) | 1
  Pt #17 Social Functioning : Visit 5 | NA — Data not collected
  Pt #17 Social Functioning : Visit 8: number analyzed (Participants) | 1
  Pt #17 Social Functioning : Visit 8 | 50
  Pt #17 Social Functioning : Visit 9: number analyzed (Participants) | 1
  Pt #17 Social Functioning : Visit 9 | 50
  Pt #17 Social Functioning : Visit 10: number analyzed (Participants) | 1
  Pt #17 Social Functioning : Visit 10 | NA — Data not collected
  Pt #17 Pain : Visit 1: number analyzed (Participants) | 1
  Pt #17 Pain : Visit 1 | 100
  Pt #17 Pain : Visit 5: number analyzed (Participants) | 1
  Pt #17 Pain : Visit 5 | NA — Data not collected
  Pt #17 Pain : Visit 8: number analyzed (Participants) | 1
  Pt #17 Pain : Visit 8 | 100
  Pt #17 Pain : Visit 9: number analyzed (Participants) | 1
  Pt #17 Pain : Visit 9 | 75
  Pt #17 Pain : Visit 10: number analyzed (Participants) | 1
  Pt #17 Pain : Visit 10 | NA — Data not collected
  Pt #17 General Health : Visit 1: number analyzed (Participants) | 1
  Pt #17 General Health : Visit 1 | 55
  Pt #17 General Health : Visit 5: number analyzed (Participants) | 1
  Pt #17 General Health : Visit 5 | NA — Data not collected
  Pt #17 General Health : Visit 8: number analyzed (Participants) | 1
  Pt #17 General Health : Visit 8 | 70
  Pt #17 General Health : Visit 9: number analyzed (Participants) | 1
  Pt #17 General Health : Visit 9 | 55
  Pt #17 General Health : Visit 10: number analyzed (Participants) | 1
  Pt #17 General Health : Visit 10 | NA — Data not collected

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each patient during treatment and in follow up for up to 18 weeks.
Arm/Group | Bortezomib
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=17)
Myocardial Infarction (Cardiac disorders) | 1
Dehydration (Gastrointestinal disorders) | 1 — Patient also will diarrhea and syncope at the time of the event
Varicella aoster virus/systemic inflammatory response (Infections and infestations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=17)
Hemoglobin (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 7
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3
Insomnia (General disorders) | 2
Sweating (diaphoresis) (General disorders) | 1
Weight gain (General disorders) | 1
Weight loss (General disorders) | 3
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other (Specify: skin lesion with some oozing) (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 1
Infection - Systemic Inflammatory Response Syndrome (Infections and infestations) | 1
Infection - pulmonary/upper respiratory - upper airway NOS (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Nose (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Pharynx (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1
Viral hepatitis (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Mood alteration - Anxiety (Nervous system disorders) | 1
Mood alteration - Depression (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 8
Syncope (fainting) (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 3
Ocular/Visual - Other (Specify, Meibomitis) (Eye disorders) | 2
Vision-blurred vision (Eye disorders) | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest Wall (Cardiac disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Flu-like syndrome (General disorders) | 3

LIMITATIONS AND CAVEATS:
The study was closed before the accrual goal of 20 evaluable patients was reached due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No